CLINICAL TRIAL: NCT02431156
Title: Retrospective Functional Assessment of Activities of Daily Living (ADL) in Patients Who Underwent Mini-monovision Correction With Bilateral Implantation of Aspheric Monofocal Intraocular Lenses
Brief Title: Functional Assessment of Activities of Daily Living (ADL) in Patients Who Underwent Mini-monovision Correction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Assistant Professor, Democritus University of Thrace
Other Study IDs: PseudoPresbADL
Record Dates: First submitted 2015-04-01; First posted 2015-04-30 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Presbyopia
Keywords: presbyopia; monovision; activities of daily living,; pseudophakic
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- monovision: Presbyopic patients that underwent mini-monovision correction with bilateral implantation of monofocal intraocular lenses. Their visual capacity in ADLs will be assessed.
  Interventions: Other: Assessment of visual capacity

INTERVENTIONS:
Other: Assessment of visual capacity — Visual capacity (VC) is variable comprised by three sub-variables: a) (DVC) Visual capacity for activities requiring distant vision, b) (IVC) Visual capacity for activities requiring intermediate vision, and c) (NVC) Visual capacity for activities requiring near vision.
  VC will be measured in a scale from 1 to 100 as the sum of the DVC, IVC and NVC

SUMMARY:
Patients who underwent mini-monovision (with bilateral myopic defocus, MM-BMD) surgery for presbyopia correction with monofocal intraocular lenses implantation are supposed to have sufficient uncorrected vision capacity for activities of daily living (ADLs) that require: a) distant vision(DV), (ie. driving), b) intermediate vision (IV), (ie. computer word processing), c) near vision (NV), (ie. book reading). Primary objectives of the study are: 1) the development of a series of tasks in a research setting that will simulate common ADLs that require DV, IV, and NV. 2) the identification of potential correlations of the tasks in the research setting with demographic, clinical and other parameters of the study participants.

DETAILED DESCRIPTION:
Patients who underwent mini-monovision (with bilateral myopic defocus, MM-BMD) surgery for presbyopia correction with monofocal intraocular lenses implantation are supposed to have sufficient uncorrected vision capacity for activities of daily living (ADLs) that require: a) distant vision(DV), (ie. driving), b) intermediate vision (IV), (ie. computer word processing), c) near vision (NV), (ie. book reading). Primary objectives of the study are: 1) the development of a series of tasks in a research setting that will simulate common ADLs that require DV, IV, and NV. 2) the identification of potential correlations of the tasks in the research setting with demographic, clinical and other parameters of the study participants

ELIGIBILITY:
Inclusion Criteria:

* Presbyopic patients that underwent mini-monovision correction with bilateral myopic defocus with monofocal intraocular lenses implantation

Exclusion Criteria:

* Glaucoma
* Corneal pathology
* Fundus pathology
* Severe neurological/mental diseases that interfere with visual acuity

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Presbyopic patients that underwent mini-monovision correction with bilateral myopic defocus with monofocal intraocular lenses implantation
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of Visual capacity (VC) | 1 year following mini-monovision correction surgery
  VC will be measured as the sum of DVC, IVC, and NVC

SECONDARY OUTCOMES:
Visual capacity for activities that require distant vision (DVC) | 1 year following mini-monovision correction surgery
  DVC score will be measured by the performance score in the following ADLs: a) walking specific pathway, 2) walking up stairs, 3) walking down stairs, 4) day-time driving simulation, 5) night-time driving simulation
Visual capacity for activities that require intermediate vision (IVC) | 1 year following mini-monovision correction surgery
  IVC score will be measured by the performance score in the following ADLs: a) reading ability of movie subtitles, b) reading ability of a predefined computer screen text, c) reading a supermarket badge
Visual capacity for activities that require near vision (NVC) | 1 year following mini-monovision correction surgery
  NVC score will be measured by the performance score in the following ADLs: a) cellular phone directory entry search, b) reading of message in a cellular phone, c) reading a medical prescription, d) reading a public phonebook

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Eye Institute Of thrace, Alexandroupoli, Evros, Greece

REFERENCES:
- [Derived] Labiris G, Ntonti P, Patsiamanidi M, Sideroudi H, Georgantzoglou K, Kozobolis VP. Evaluation of activities of daily living following pseudophakic presbyopic correction. Eye Vis (Lond). 2017 Jan 19;4:2. doi: 10.1186/s40662-016-0067-1. eCollection 2017. PMID 28116335